CLINICAL TRIAL: NCT07335523
Title: A Phase 2 Treatment Withdrawal Clinical Trial of a Bicarbonate-Buffered, Enteric-Coated Pancreatic Enzyme Supplement for the Management of Steatorrhea in Children and Young Adults With Alagille Syndrome After Liver Transplantation
Brief Title: Management of Steatorrhea in Children and Young Adults With Alagille Syndrome After Liver Transplantation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Digestive Care, Inc. (Industry)
Collaborators: Alagille Syndrome Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102824-001
Record Dates: First submitted 2026-01-08; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Steatorrhea
Keywords: Alagille Syndrome; steatorrhea; liver transplant; fecal fat; Pertzye; coefficient of fat; exocrine pancreatic insufficiency
MeSH Terms: conditions — Steatorrhea; Alagille Syndrome; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Intervention Model Description: Treatment withdrawal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PERTZYE (Experimental): PERTZYE (pancrelipase) delayed-release capsules, for oral administration
  Interventions: Drug: Pertzye

INTERVENTIONS:
Drug: Pertzye — PERTZYE (pancrelipase) delayed-release capsules

SUMMARY:
The goal of this clinical trial is to learn if PERTZYE® works to treat steatorrhea in children and adults with Alagille Syndrome (ALGS) post liver transplant. It will also learn about the safety of PERTZYE®. The main questions it aims to answer are:

* Does PERTZYE improve dietary fat absorption?
* Does PERTZYE improve stool frequency and consistency?
* Does PERTZYE improve abdominal signs and symptoms?
* What medical problems do participants have when taking PERTZYE? Researchers will compare the results when participants are taking and stop taking PERTZYE.

During the study, participants will:

* Consume a high fat diet
* Take PERTZYE every day with meals and snacks for up to 4 weeks
* Have scheduled checkups by phone or video by clinical staff
* Keep a diary of their symptoms and PERTZYE dosing
* Collect stool for laboratory testing

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ages 7-50 years inclusive.
* Confirmed diagnosis of ALGS
* Status post OLT due to ALGS complications.
* Participants currently managed with pancreatic enzyme products (PEPs) are allowed pending discontinuation of PEPs for 5 days prior to beginning the 72-hour stool collections. Participants must discontinue PEPs for the entire study period until completion.
* Agree to adhere to a high fat diet at least 2 days prior to and during the 72-hour stool collections and monitor dietary consumption through the use of a diet diary.
* Presence of steatorrhea confirmed by baseline CFA ≤ 90%.
* Have a consistent caregiver for the duration of the study if applicable for enrollment of a child.
* Capable of giving written informed consent and assent (if age appropriate).

Exclusion Criteria:

* Surgical disruption of the enterohepatic circulation (e.g., biliary diversion).
* Diets high in medium-chain triglyceride (MCT) oil.
* Use of bile acids, bile acid uptake inhibitors, lipid-binding resins, synthetic fat substitutes (e.g. Olestra), and diaper rash ointments (note that H2 antagonists and proton pump inhibitors [PPIs] are permitted if on a stable and consistent regimen throughout the duration of the study).
* History or presence of other concomitant liver diseases such as liver transplant rejection with cholestasis, hepatitis B or C virus infection, HIV, primary sclerosing cholangitis (PSC), alcoholic liver disease, autoimmune hepatitis, metabolic-associated fatty liver disease (MASLD)/non-alcoholic steatohepatitis (NASH) or significant chronic allograft rejection.
* Currently pregnant or breastfeeding.
* Cancers except for in situ carcinoma or cancers treated at least 5 years prior to screening with no evidence of recurrence.
* Participation in a clinical trial and received an investigational product within the last 30 days.
* Use of anti-diarrheal, anti-spasmodic, and/or cathartic laxatives. Change in osmotic laxatives within the past 3 months.

Ages: 7 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in dietary fat absorption | End of the 4 week treatment period
  Improvement in dietary fat absorption is measured by calculating the percent of fat absorption (0-100%). Higher percentage of fat absorption indicates improvement.

IPD SHARING:
Plan to Share IPD: No